CLINICAL TRIAL: NCT03315767
Title: Prospective Evaluation of Non-invasive ARFI-elastography of Liver and Spleen and Portal Flow Measurement in Comparison With Invasive HVPG (Hepatic Venous Pressure Gradient)-Measurement for Patients With Portal Hypertension.
Brief Title: Spleen-ARFI-assisted-Portal-Hypertension-Evaluation-Study (SAPHES)
Acronym: SAPHES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Thomas Seufferlein, Head of Department Internal Medicine I, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SAPHES
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Hypertension, Portal
Keywords: HVPG; portal hypertension; ARFI; portal vein flow; advanced liver chronic disease (ACLD)
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cirrhosis patients (Other): ARFI-elastography and portal vein flow measurement: Liver and spleen of patients with a scheduled HVPG-investigation will be examined by an ARFI-elastography-investigation. Additionally the portal vein flow will be assessed.
  This examination will be done at d0 before the start of beta-blocker-administration and repeated as monitoring for portal hypertension treated by beta-blocker after 6 and 12 weeks, respectively.
  HVPG-measurement: HVPG-values will be assessed at d0, after 6 and after 12 Weeks, respectively.
  Interventions: Diagnostic Test: ARFI-elastography and portal vein flow measurement; Diagnostic Test: HVPG-measurement

INTERVENTIONS:
Diagnostic Test: ARFI-elastography and portal vein flow measurement — Liver and spleen-elastography assessed by ARFI-technique and the portal vein flow value-assessment by ultrasound investigation.
Diagnostic Test: HVPG-measurement — Evaluation of Portal Hypertension by HVPG-measurement

SUMMARY:
This study evaluates correlation in changes of HVPG-pressure values and stiffness values (ARFI) for spleen and liver and flow-volume values in Portal vein in patients with liver cirrhosis/Portal Hypertension, respectively, after new-admission of beta-blocker therapy.

DETAILED DESCRIPTION:
Portal Hypertension is the most important risk factor for development of liver cirrhosis-linked complications (e.g. ascites, variceal bleeding, hepatocellular carcinoma, etc.). The invasive HVPG-technique is the standard-of-care Investigation for Evaluation of Portal Hypertension. Administration of Beta-Blocker-therapy results in dropping of the elevated Portal vein pressure values so Overall-survival rate and incidence of liver-cirrhosis-linked complications can be ameliorated. Ultrasound-based Investigation of liver and Spleen-stiffness and of portal-vein-flow-volume, respectively, are the non-invasive methods for Evaluation of Portal Hypertension. But the cut-off values for detection of significant Portal Hypertension by the ultrasound investigation strongly vary depending on the study performed. This study evaluates the changes in ARFI-assisted elastography measurements of liver and spleen and in portal vein flow values, respectively, compared with the recorded Delta in invasive hepatic vein pressure gradient (HVPG)-values for patients with portal hypertension and new administered beta-blocker-therapy. The aim of this study is to evaluate value drop in liver- and Spleen-stiffness and portal-vein-flow required in corelation to a significant drop in HVPG-pressure after new-administered beta-blocker therapy.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis
* portal hypertension
* indication to beta-blocker-therapy

Exclusion Criteria:

* contraindication to beta-blocker-therapy
* HVPG-measurement not feasible
* portal vein thrombosis
* hematologic underlying disease as the source for enlarged/stiff spleen or liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in ARFI-elastography value for spleen due to beta-blocker therapy | 6 and 12 weeks
  ARFI-elastography: measured in m/s

SECONDARY OUTCOMES:
Correlation between changes in HVPG-values and ARFI-elastography values for liver | 6 and 12 weeks
  HVPG-values: measured in mmHg; ARFI-elastography: measured in m/s
Correlation between changes in HVPG-values and ARFI-elastography values for spleen | 6 and 12 weeks
  HVPG-values: measured in mmHg; ARFI-elastography: measured in m/s
Correlation between changes in HVPG-values and portal vein flow measurements | 6 and 12 weeks
  HVPG-values: measured in mmHg; Portal vein flow: measured in cm/s
Correlation between changes in grade of esophageal varices and HVPG-values | 12 weeks
  esophageal varices: modified Poquet classification; HVPG-values: measured in mmHg
Correlation between changes in grade of esophageal varices and ARFI-values for liver | 12 weeks
  esophageal varices: modified Poquet classification; ARFI-elastography: measured in m/s
Correlation between changes in grade of esophageal varices and ARFI-values for spleen | 12 weeks
  esophageal varices: modified Poquet classification; ARFI-elastography: measured in m/s
Correlation between changes in grade of esophageal varices and Portal vein flow | 12 weeks
  Portal vein flow: measured in cm/s; esophageal varices: modified Poquet classification
Change in ARFI-elastography value for liver due to beta-blocker therapy | 6 and 12 weeks
  ARFI-elastography: measured in m/s
Change in portal vein flow value due to beta-blocker therapy | 6 and 12 weeks
  Portal vein flow: measured in cm/s

CONTACTS AND LOCATIONS:
Overall Officials: Eugen Zizer, MD, Principal Investigator — University of Ulm
Locations (1):
- Universitätsklinikum Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Binzberger A, Hanle M, Pfahler M, Kratzer W, Seufferlein T, Zizer E. Spleen and Liver Stiffness Evaluation by ARFI Imaging: A Reliable Tool for a Short-Term Monitoring of Portal Hypertension? Int J Hepatol. 2022 Sep 9;2022:7384144. doi: 10.1155/2022/7384144. eCollection 2022. PMID 36117519